CLINICAL TRIAL: NCT02165215
Title: Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy (Maintenance of Remission) and Safety of Etrolizumab Compared With Placebo in Patients With Moderate to Severe Active Ulcerative Colitis Who Are Naive to TNF Inhibitors
Brief Title: A Study of the Efficacy and Safety of Etrolizumab Treatment in Maintenance of Disease Remission in Ulcerative Colitis (UC) Participants Who Are Naive to Tumor Necrosis Factor (TNF) Inhibitors
Acronym: LAUREL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA29102; 2013-004280-31 (EudraCT Number)
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Open-Label Induction Phase: Etrolizumab (Experimental): All participants will receive treatment with open-label etrolizumab 105 milligrams (mg) subcutaneous (SC) injection once every 4 weeks (Q4W) up to Week 10.
  Interventions: Drug: Etrolizumab
- Double-Blind Maintenance Phase: Etrolizumab (Experimental): Participants who achieved a clinical response at Week 10 during the induction phase and randomized to this arm for the double-blind maintenance phase will receive etrolizumab 105 mg SC injection Q4W from Week 12 up to Week 62.
  Interventions: Drug: Etrolizumab
- Double-Blind Maintenance Phase: Placebo (Placebo Comparator): Participants who achieved a clinical response at Week 10 during the induction phase and randomized to this arm for the double-blind maintenance phase will receive placebo (matched to etrolizumab) SC injection Q4W from Week 12 up to Week 62.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etrolizumab — Participants will receive 105 mg etrolizumab SC injection Q4W.
  Other Names: RG7413; RO5490261; PRO145223; rhuMAb Beta7
  Arms: Double-Blind Maintenance Phase: Etrolizumab; Open-Label Induction Phase: Etrolizumab
Drug: Placebo — Participants will receive placebo (matched to etrolizumab) SC injection Q4W.
  Arms: Double-Blind Maintenance Phase: Placebo

SUMMARY:
This Phase III, randomized, double-blind, parallel-grouped, placebo-controlled, multicenter study will investigate the efficacy and safety of etrolizumab in maintenance of remission in participants with moderately to severely active UC who are naive to TNF inhibitors and refractory to or intolerant of prior immunosuppressant and/or corticosteroid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis (UC) established at least 3 months prior to Day 1 by clinical and endoscopic evidence
* Moderately to severely active UC as determined by an MCS of 6-12 with an endoscopic subscore greater than or equal to (≥)2 as determined by the central reading procedure (endoscopy to be performed 4-16 days prior to Day 1), a rectal bleeding subscore ≥1, and a stool frequency subscore ≥1 during the screening period (prior to Day 1)
* Evidence of UC extending a minimum of 20 centimeters (cm) from the anal verge as determined by baseline endoscopy (flexible sigmoidoscopy or colonoscopy) performed during screening, 4-16 days prior to Day 1
* Naive to treatment with any anti-TNF therapy
* Participants must have had an inadequate response, loss of response, or intolerance to prior corticosteroid and/or immunosuppressant treatment
* Background regimen for UC may include oral 5-aminosalicylate (5-ASA), oral corticosteroids, budesonide, probiotics, azathioprine (AZA), 6-mercaptopurine (6-MP), or methotrexate (MTX) if doses have been stable during the screening period
* Use of highly effective contraception
* Must have received a colonoscopy within the past year or be willing to undergo a colonoscopy in lieu of a flexible sigmoidoscopy at screening

Exclusion Criteria:

* A history of or current conditions and diseases affecting the digestive tract, such as indeterminate colitis, suspicion of ischemic colitis, radiation colitis, or microscopic colitis, Crohn's disease, fistulas or abdominal abscesses, colonic mucosal dysplasia, intestinal obstruction, toxic megacolon, or unremoved adenomatous colonic polyps
* Prior or planned surgery for UC
* Past or present ileostomy or colostomy
* Any prior treatment with etrolizumab or other anti-integrin agents (including natalizumab, vedolizumab, and efalizumab) as stated in the protocol
* Any prior treatment with anti-adhesion molecules (such as mucosal addressin cell adhesion molecule [MAdCAM-1])
* Any prior treatment with rituximab
* Any treatment with tofacitinib during screening
* Cogenital or acquired immune deficiency, chronic hepatitis B or C infection, human immunodeficiency virus (HIV) positive, or history of tuberculosis (active or latent)
* Evidence of or treatment for Clostridium difficile within 60 days prior to Day 1 or other intestinal pathogens within 30 days prior to Day 1
* History of recurrent opportunistic infections and/or severe disseminated viral infections
* History of organ transplant
* Any major episode of infection requiring treatment with intravenous (IV) antibiotics within 8 weeks prior to screening or oral antibiotics within 4 weeks prior to screening
* Received a live attenuated vaccine within 4 weeks prior to Day 1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (104):
- United States (33):
  - University of California, Irvine Medical Center, Orange, California
  - Clinical Applications Laboratories, Inc., San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Ventura Clinical Trials, Ventura, California
  - Peak Gastroenterology Associates; Gastroenterology, Colorado Springs, Colorado
  - Clinical Research of the Rockies, Lafayette, Colorado
  - West Central Gastroenterology d/b/a Gastro Florida, Clearwater, Florida
  - Regenerate Clinical Trials, Miami, Florida
  - IMIC, Inc, Miami Beach, Florida
  - Advanced Research Institute, Inc., Trinity, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Northwestern University-Feinberg School of Medicine; Division of Gastroenterology and Hepatology, Chicago, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Aquiant Research, New Albany, Indiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Center for Digestive Health, Troy, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ehrhardt Clinical Research, LLC, Belton, Missouri
  - Manhattan Clinical Research, New York, New York
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - UNC at Chapel Hill - Dpt of Family Medicine; Center for Functional GI and Motility Disorders, Chapel Hill, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Texas Digestive Disease Consultants - Dallas, Dallas, Texas
  - Texas Digestive Disease Consultants - Southlake, Southlake, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - Ericksen Research and Development, Clinton, Utah
  - University of Utah School of Medicine, Salt Lake City, Utah
  - McGuire Research Institute; Gastroenterology, Richmond, Virginia
  - Northwest Gastroenterology Associates, Bellevue, Washington
- Brazil (8):
  - Hospital Universitario Walter Cantidio - UFC, Fortaleza, Ceará
  - Centro Digestivo de Curitiba, Curitiba, Paraná
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - CECIP - Centro de Estudos Clínicos do Interior Paulista, Jaú, São Paulo
  - Pesquisare Saúde Sociedade Simples, Santo André, São Paulo
  - Hospital Estadual Mario Covas, Santo André, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Hospital do Servidor Público Estadual/HSPE-SP, São Paulo, São Paulo
- Canada (6):
  - Pacific Gastroenterology Associates, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre; Gastroenterology Research, Halifax, Nova Scotia
  - LHSC - University Hospital; Movement Disorders Program, London, Ontario
  - London Health Sciences Centre Victoria Hospital; Research Pharmacy, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Digestive Disease Associates, Vaughan, Ontario
- Czechia (3):
  - Fakultni nemocnice u sv. Anny v Brne; I.Interni kardioangiologicka klinika, Brno
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Nemocnice Na Bulovce, Prague
- Denmark (2):
  - Alborg Universitets Hospital, Aalborg
  - Herlev og Gentofte Hospital, Herlev
- Germany (8):
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Berufsgenossenschaftliches Universitaetsklinikum Bergmannsheil GmbH, Bochum
  - Ärztezentrum Ellwangen; Gemeinschaftspraxis, Ellwangen
  - Klinik Johann Wolfgang von Goethe Uni, Frankfurt
  - Medizinische Hochschule Hannover; Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Hanover
  - Universitaetsklinikum Jena; Apotheke des Uniersitätsklinikums Jena, Jena
  - Medizinisches Zentrum Klinikum Lueneburg, Lüneburg
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
- Hungary (5):
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Pannónia Klinika Magánorvosi, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz, Szentes
- India (13):
  - Osmania General Hospital, Hyderabad, Andhra Pradesh
  - Deccan College of Medical Sciences and Allied Hospitals, Hyderabad, Andhra Pradesh
  - Shree Giriraj Multispeciality Hospital, Rajkot, Gujarat
  - Nirmal Hospital, Surat, Gujarat
  - K.L.E. Society's Dr. Prabhakar Kore Hospital and Medical Research Centre, Belagavi, Karnataka
  - M. S. Ramaiah Medical College and Hospital, Bengaluru, Karnataka
  - Midas institute of Gastroenterology, Nagpur, Maharashtra
  - Pushpawati Singhania Research Institute, New Delhi, National Capital Territory of Delhi
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - S. R. Kalla Memorial General Hospital, Jaipur
  - Kasturba Medical College & Hospital, Mangalore
  - Ruby Hall Clinic, Pune
  - King Edward Memorial Hospital Research Centre, Pune
- Israel (5):
  - Assaf Harofeh Medical Center, Beer Yaacov
  - Bnei Zion Medical Center; Department of Internal Medicine B, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Holy Family Hospital, Nazareth
- Italy (4):
  - Ospedale Sandro Pertini, Rome, Lazio
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia, Lombardy
  - Ospedale di Circolo; Neuropsichiatria Infantile, Rho, Lombardy
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo, Sicily
- Mexico (3):
  - Centro Regiomontano de Estudios Clínicos Roma S.C., Monterrey, Nuevo León
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Phylasis Clinicas Research S de RL de CV, Estado de México
- Poland (2):
  - Zespó Przychodni Specjalistycznych PRIMA, Warsaw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
- Slovakia (2):
  - Fakultna nemocnica Nitra, Nitra
  - Endomed, s.r.o., Vranov nad Topľou
- South Africa (2):
  - Dr JP Wright Practice, Cape Town
  - Emmed Research, Pretoria
- Ukraine (8):
  - CI of SRC Sumy RCH Dept of Rheumatology Sumy SU MI, Sumy, Kharkiv Governorate
  - CI of Kyiv RC Kyiv Regional Clinical Hospital, Kyiv, KIEV Governorate
  - Lviv Regional Clinical Hospital, Lviv, KIEV Governorate
  - A.Novak Transcarpathian Regional Clinical Hospital, Uzhhorod, KIEV Governorate
  - Odessa regional clinical Hospital, Odesa
  - M.V. Sklifosovskyi Poltava RCH Dept of Gastroenterology HSEIU UMSA, Poltava
  - SI Divisional Clinical Hospital of Uzhgorod Station of ST&BA LZ Dep of Therapy SHEI Uzhgorod NU, Uzhhorod
  - M.I. Pyrogov VRCH Dept of Gastroenterology M.I. Pyrogov VNMU, Vinnytsia

REFERENCES:
- [Derived] Vermeire S, Lakatos PL, Ritter T, Hanauer S, Bressler B, Khanna R, Isaacs K, Shah S, Kadva A, Tyrrell H, Oh YS, Tole S, Chai A, Pulley J, Eden C, Zhang W, Feagan BG; LAUREL Study Group. Etrolizumab for maintenance therapy in patients with moderately to severely active ulcerative colitis (LAUREL): a randomised, placebo-controlled, double-blind, phase 3 study. Lancet Gastroenterol Hepatol. 2022 Jan;7(1):28-37. doi: 10.1016/S2468-1253(21)00295-8. Epub 2021 Nov 17. PMID 34798037
- [Derived] Sandborn WJ, Vermeire S, Tyrrell H, Hassanali A, Lacey S, Tole S, Tatro AR; Etrolizumab Global Steering Committee. Etrolizumab for the Treatment of Ulcerative Colitis and Crohn's Disease: An Overview of the Phase 3 Clinical Program. Adv Ther. 2020 Jul;37(7):3417-3431. doi: 10.1007/s12325-020-01366-2. Epub 2020 May 22. PMID 32445184

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 359 participants were enrolled into the OLI phase of the study. A total of 210 participants were randomized into the Maintenance phase and received either Etrolizumab or Placebo.
Period: Induction Phase
Arm/Group | Open-Label Induction Phase: Etrolizumab | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Started | 359 | 0 | 0
Dosed | 358 | 0 | 0
Completed | 336 | 0 | 0
Not Completed | 23 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Non-Compliance | 2 | 0 | 0
Not completed — Lost to Follow-up | 6 | 0 | 0
Period: Maintenance Phase
Arm/Group | Open-Label Induction Phase: Etrolizumab | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Started | 0 | 108 | 106
Dosed | 0 | 108 | 102
Completed | 0 | 96 | 101
Not Completed | 0 | 12 | 5
Not completed — Withdrawal by Subject | 0 | 7 | 3
Not completed — Multiple reasons | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-Label Induction Phase: Etrolizumab | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo | Total
Number analyzed (Participants) | 359 | 108 | 106 | 573
Age, Continuous [Mean (Standard Deviation); unit: years] — Maintenance Phase Population: Participants in the Maintenance Phase of the study
  years
    number analyzed (Participants) | 0 | 108 | 106 | 214
    (all) |  | 38.3 (13.7) | 39.2 (13.5) | 38.7 (13.6)
Age, Continuous [Mean (Standard Deviation); unit: years] — Induction Phase Population: Participants in the Induction Phase of the study
  years
    number analyzed (Participants) | 359 | 0 | 0 | 359
    (all) | 39.2 (13.9) |  |  | 39.2 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Maintenance Phase Population: Participants in the Maintenance Phase of the study
  Participants
    number analyzed (Participants) | 0 | 108 | 106 | 214
    Female |  | 48 | 54 | 102
    Male |  | 60 | 52 | 112
Sex: Female, Male [Count of Participants; unit: Participants] — Induction Phase Population: Participants in the Induction Phase of the study
  Participants
    number analyzed (Participants) | 359 | 0 | 0 | 359
    Female | 156 |  |  | 156
    Male | 203 |  |  | 203
Race (NIH/OMB) [Count of Participants; unit: Participants] — Maintenance Phase Population: Participants in the Maintenance Phase of the study
  Participants
    number analyzed (Participants) | 0 | 108 | 106 | 214
    American Indian or Alaska Native |  | 2 | 2 | 4
    Asian |  | 21 | 13 | 34
    Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0
    Black or African American |  | 2 | 6 | 8
    White |  | 79 | 78 | 157
    More than one race |  | 0 | 0 | 0
    Unknown or Not Reported |  | 4 | 7 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants] — Induction Phase Population: Participants in the Induction Phase of the study
  Participants
    number analyzed (Participants) | 359 | 0 | 0 | 359
    American Indian or Alaska Native | 5 |  |  | 5
    Asian | 58 |  |  | 58
    Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
    Black or African American | 13 |  |  | 13
    White | 269 |  |  | 269
    More than one race | 0 |  |  | 0
    Unknown or Not Reported | 14 |  |  | 14

OUTCOME MEASURES:

1. Primary Outcome: Maintenance Phase: Percentage of Participants in Remission at Week 62 Among Randomized Participants With a Clinical Response at Week 10, as Determined by the Mayo Clinic Score (MCS)
Description: MCS is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy, and physician's global assessment.
  Clinical Response is MCS with ≥3-point decrease and 30% reduction from baseline as well as ≥1-point decrease in rectal bleeding subscore or an absolute rectal bleeding score of 0 or 1.
  Remission is MCS ≤2 with individual subscores ≤1 and a rectal bleeding subscore of 0.
Time Frame: Week 62
Population: Participants in the Maintenance phase of the study that received an intervention
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 108 | 102
percentage of participants | 29.6 | 20.6
Statistical Analysis 1: Comparison: Double-Blind Maintenance Phase: Etrolizumab vs Double-Blind Maintenance Phase: Placebo; Test type: Superiority; p = 0.1942, Cochran-Mantel-Haenszel; Adjusted difference in response rates = 7.7, 95% CI 2-sided [-4.2 to 19.2]

2. Secondary Outcome: Maintenance Phase: Percentage of Participants Who Maintained Clinical Remission at Week 62 Among Randomized Participants in Clinical Remission at Week 10, as Determined by the MCS
Description: MCS is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy, and physician's global assessment.
  Clinical Remission is MCS ≤2 with individual subscores ≤1.
Time Frame: Week 62
Population: Participants in the Maintenance phase of the study that had Clinical Remission at Week 10
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 45 | 44
percentage of participants | 44.4 | 27.3
Statistical Analysis 1: Comparison: Double-Blind Maintenance Phase: Etrolizumab vs Double-Blind Maintenance Phase: Placebo; Test type: Superiority; p = 0.1524, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted difference in remission rates = 14.6, 95% CI 2-sided [-5.55 to 33.15]

3. Secondary Outcome: Maintenance Phase: Percentage of Participants in Clinical Remission at Week 62, as Determined by the MCS
Description: as for outcome 2
Time Frame: Week 62
Population: Participants in the Maintenance phase of the study that received an intervention
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 108 | 102
percentage of participants | 30.6 | 20.6
Statistical Analysis 1: Comparison: Double-Blind Maintenance Phase: Etrolizumab vs Double-Blind Maintenance Phase: Placebo; Test type: Superiority; p = 0.1466, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted difference in remission rates = 8.7, 95% CI 2-sided [-3.26 to 20.21]

4. Secondary Outcome: Maintenance Phase: Percentage of Participants in Remission at Week 62 Among Randomized Participants in Remission at Week 10, as Determined by the MCS
Description: MCS is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy, and physician's global assessment.
  Remission is MCS ≤2 with individual subscores ≤1 and a rectal bleeding subscore of 0.
Time Frame: Week 62
Population: Participants in the Maintenance phase of the study that had Remission at Week 10
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 40 | 41
percentage of participants | 40.0 | 26.8
Statistical Analysis 1: Comparison: Double-Blind Maintenance Phase: Etrolizumab vs Double-Blind Maintenance Phase: Placebo; Test type: Superiority; p = 0.3083, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted difference in remission rates = 10.9, 95% CI [-9.72 to 30.49]

5. Secondary Outcome: Maintenance Phase: Percentage of Participants With Improvement From Baseline in Endoscopic Appearance of the Mucosa at Week 62, as Determined by the MCS Endoscopic Subscore
Description: MCS is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy, and physician's global assessment.
  Improvement in endoscopic appearance of the mucosa is Endoscopy subscore ≤1.
Time Frame: Baseline, Week 62
Population: Participants in the Maintenance phase of the study that received an intervention
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 108 | 102
percentage of participants | 38.0 | 22.5
Statistical Analysis 1: Comparison: Double-Blind Maintenance Phase: Etrolizumab vs Double-Blind Maintenance Phase: Placebo; Test type: Superiority; p = 0.0235, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted difference in response rates = 14.4, 95% CI 2-sided [1.84 to 26.28]

6. Secondary Outcome: Maintenance Phase: Percentage of Participants With Endoscopic Remission at Week 62, as Determined by the MCS Endoscopic Subscore
Description: MCS is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy, and physician's global assessment.
  Endoscopic Remission is Endoscopy subscore = 0.
Time Frame: Week 62
Population: Participants in the Maintenance phase of the study that received an intervention
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 108 | 102
percentage of participants | 30.6 | 16.7
Statistical Analysis 1: Comparison: Double-Blind Maintenance Phase: Etrolizumab vs Double-Blind Maintenance Phase: Placebo; Test type: Superiority; p = 0.0293, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted difference in remission rates = 12.8, 95% CI [1.13 to 23.89]

7. Secondary Outcome: Maintenance Phase: Percentage of Participants With Histologic Remission at Week 62, as Determined by the Nancy Histological Index
Description: Nancy Histological Index (NHI) is a 5-level classification ranging from grade 0 (No histologically significant disease) to grade 4 (severely active disease). Histologic remission is defined as a Nancy histological index of 0 or 1.
Time Frame: Week 62
Population: Participants in the Maintenance phase of the study that were evaluated using the Nancy histological index (enrolled after the latest protocol amendment)
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 85 | 78
percentage of participants | 42.4 | 21.8
Statistical Analysis 1: Comparison: Double-Blind Maintenance Phase: Etrolizumab vs Double-Blind Maintenance Phase: Placebo; Test type: Superiority; p = 0.0075, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted difference in remission rates = 19.8, 95% CI 2-sided [5.16 to 33.11]

8. Secondary Outcome: Maintenance Phase: Percentage of Participants With Corticosteroid-Free Clinical Remission at Week 62 Among Participants Who Were Receiving Corticosteroids at Baseline, as Determined by the MCS
Description: as for outcome 2
Time Frame: Baseline, Week 62
Population: Participants in the Maintenance phase of the study receiving Corticosteroids at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 55 | 50
percentage of participants | 18.2 | 8.0
Statistical Analysis 1: Comparison: Double-Blind Maintenance Phase: Etrolizumab vs Double-Blind Maintenance Phase: Placebo; Test type: Superiority; p = 0.1415, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted difference in remission rates = 9.9, 95% CI [-4.47 to 23.13]

9. Secondary Outcome: Maintenance Phase: Percentage of Participants With Corticosteroid-Free Remission at Week 62 Among Participants Who Were Receiving Corticosteroids at Baseline, as Determined by the MCS
Description: as for outcome 4
Time Frame: Baseline, Week 62
Population: Participants in the Maintenance phase of the study receiving Corticosteroids at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 55 | 50
percentage of participants | 18.2 | 8.0
Statistical Analysis 1: Comparison: Double-Blind Maintenance Phase: Etrolizumab vs Double-Blind Maintenance Phase: Placebo; Test type: Superiority; p = 0.1415, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted difference in remission rates = 9.9, 95% CI [-4.47 to 23.13]

10. Secondary Outcome: Maintenance Phase: Change From Baseline to Week 62 in UC Bowel Movement Signs and Symptoms, as Assessed by the Ulcerative Colitis Patient-Reported Outcome Signs and Symptoms (UC-PRO/SS) Questionnaire
Description: The UC-PRO questionnaire is collected in the e-diary and completed by participants for at least 9-12 consecutive days prior to a study visit. The UC-PRO is being reported in three domains; two domains are key endpoints and reported as UC-PRO Signs and Symptoms (UC-PRO/SS).
  The bowel domain score ranges from 0-27, with a higher score indicating a worse disease state.
Time Frame: Baseline, Week 62
Population: Participants in the Maintenance phase of the study that completed a baseline and at least 1 post-baseline questionnaire
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 68 | 73
score on a scale | -9.6 (0.8) | -6.7 (0.9)
Statistical Analysis 1: Comparison: Double-Blind Maintenance Phase: Etrolizumab vs Double-Blind Maintenance Phase: Placebo; Test type: Superiority; p = 0.0266, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Difference in Least Square Means = -2.8, 95% CI 2-sided [-5.3 to -0.4]

11. Secondary Outcome: Maintenance Phase: Change From Baseline to Week 62 in UC Functional Symptoms, as Assessed by the UC-PRO/SS Questionnaire
Description: The UC-PRO questionnaire is collected in the e-diary and completed by participants for at least 9-12 consecutive days prior to a study visit. The UC-PRO is being reported in three domains; two domains are key endpoints and reported as UC-PRO Signs and Symptoms (UC-PRO/SS).
  The functional domain score ranges from 0-12, with a higher score indicating a worse disease state.
Time Frame: Baseline, Week 62
Population: Participants in the Maintenance phase of the study that completed a baseline and at least 1 post-baseline questionnaire
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 68 | 73
score on a scale | -3.0 (0.3) | -1.8 (0.4)
Statistical Analysis 1: Comparison: Double-Blind Maintenance Phase: Etrolizumab vs Double-Blind Maintenance Phase: Placebo; Test type: Superiority; p = 0.0175, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Difference in Least Square Means = -1.2, 95% CI 2-sided [-2.2 to -0.2]

12. Secondary Outcome: Maintenance Phase: Change From Baseline to Week 62 in Health-Related Quality of Life, as Assessed by the Overall Score of the Inflammatory Bowel Disease Questionnaire (IBDQ)
Description: The IBDQ is used to assess participant's health-related quality of life (QOL). The 32-item questionnaire contains four domains: bowel symptoms (10 items), systemic symptoms (5 items), emotional function (12 items), and social function (5 items). The items are scored on a 7-point Likert scale with a higher score indicating better health-related QOL.
  IBDQ score is a total score summed up from across all 32 questions on the questionnaire. The score can range from 32-224 and the higher score indicates a better quality of life.
Time Frame: Baseline, Week 62
Population: Participants in the Maintenance phase of the study that received an intervention
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 108 | 102
scores on a scale | 66.9 (3.39) | 64.8 (3.45)
Statistical Analysis 1: Comparison: Double-Blind Maintenance Phase: Etrolizumab vs Double-Blind Maintenance Phase: Placebo; Test type: Superiority; p = 0.6331, ANCOVA — p-value has not been adjusted for multiplicity; Difference in Adjusted Mean = 2.1, 95% CI 2-sided [-6.6 to 10.8]

13. Secondary Outcome: Number of Participants With at Least One Adverse Event by Severity, According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v4.0)
Description: All adverse events (AEs) were graded for severity using the NCI-CTCAE v4.0. Any AE not specifically listed was assessed per the following 5 grades: Grade 1 = mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated. Grade 2 = moderate; minimal, local, or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living. Grade 3 = severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living. Grade 4 = life-threatening consequences or urgent intervention indicated. Grade 5 = death related to AE. Not all grades are appropriate for all AEs; some AEs have fewer than 5 options. The terms "severe" and "serious" are not synonymous and are independently assessed for each AE. Multiple occurrences of AEs were counted only once per participant at the highest (worst) grade.
Time Frame: From Baseline up to Week 74
Population: All participants that received an intervention
Measure: Number; unit: participants
Arm/Group | Open-Label Induction Phase: Etrolizumab | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 358 | 108 | 102
participants
  Grade 1 | 95 | 24 | 23
  Grade 2 | 58 | 30 | 44
  Grade 3 | 24 | 14 | 15
  Grade 4 | 3 | 2 | 0
  Grade 5 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Adverse Events Leading to Study Drug Discontinuation
Time Frame: From Baseline up to Week 74
Population: All participants that received an intervention
Measure: Number; unit: participants
Arm/Group | Open-Label Induction Phase: Etrolizumab | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 358 | 108 | 102
participants | 9 | 5 | 9

15. Secondary Outcome: Number of Participants With Serious Infection-Related Adverse Events
Time Frame: From Baseline up to Week 74
Population: All participants that received an intervention
Measure: Number; unit: participants
Arm/Group | Open-Label Induction Phase: Etrolizumab | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 358 | 108 | 102
participants | 6 | 2 | 2

16. Secondary Outcome: Number of Participants With Infection-Related Adverse Events by Severity, According to NCI-CTCAE v4.0
Description: as for outcome 13
Time Frame: From Baseline up to Week 74
Population: All participants that received an intervention
Measure: Number; unit: participants
Arm/Group | Open-Label Induction Phase: Etrolizumab | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 358 | 108 | 102
participants
  Grade 1 | 39 | 18 | 22
  Grade 2 | 21 | 17 | 10
  Grade 3 | 6 | 1 | 2
  Grade 4 | 0 | 1 | 0
  Grade 5 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Injection-Site Reactions by Severity, According to NCI-CTCAE v4.0
Description: as for outcome 13
Time Frame: From Baseline up to Week 74
Population: All participants that received an intervention
Measure: Number; unit: participants
Arm/Group | Open-Label Induction Phase: Etrolizumab | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 358 | 108 | 102
participants
  Grade 1 | 8 | 4 | 3
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Hypersensitivity Reaction Events by Severity, According to NCI-CTCAE v4.0
Description: as for outcome 13
Time Frame: From Baseline up to Week 74
Population: All participants that received an intervention
Measure: Number; unit: participants
Arm/Group | Open-Label Induction Phase: Etrolizumab | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 358 | 108 | 102
participants
  Grade 1 | 0 | 0 | 0
  Grade 2 | 1 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Malignancies
Time Frame: From Baseline up to Week 74
Population: All participants that received an intervention
Measure: Number; unit: participants
Arm/Group | Open-Label Induction Phase: Etrolizumab | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 358 | 108 | 102
participants | 0 | 2 | 1

20. Secondary Outcome: Number of Participants With Anti-Therapeutic Antibodies (ATAs) to Etrolizumab
Time Frame: Baseline, Weeks 4, 12, 24, 44, and 62, and and Early Termination/End of Safety Follow-Up (up to Week 74)
Population: Participants who received at least one dose of study treatment and had at least one baseline or post-baseline ATA result from at least one sample.
Measure: Number; unit: participants
Arm/Group | Open-Label Induction Phase: Etrolizumab | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 337 | 108 | 102
participants | 62 | 35 | 33

21. Secondary Outcome: Maintenance Phase: Etrolizumab Serum Trough Concentration (for Arms/Timepoints Above LLOQ)
Description: As per protocol, the timepoints for each arm where more than a third of the samples were above the lower limit of quantitation (LLOQ), full summary statistics (Mean and Standard Deviation) were reported. For timepoints below the LLOQ, only the Median and Max were reported as a separate outcome measure below.
Time Frame: Pre-dose (0 hour) at Baseline and Weeks 12, 24, 44, and 62
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (μg/mL)
Arm/Group | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 105 | 100
micrograms per millilitre (μg/mL)
  Week 12 | 7.66 (4.21) | 7.63 (3.67)
  Week 24: number analyzed (Participants) | 93 | 0
  Week 24 | 10 (4.86) |
  Week 44: number analyzed (Participants) | 84 | 0
  Week 44 | 10 (4.88) |
  Week 62: number analyzed (Participants) | 75 | 0
  Week 62 | 15.4 (7.46) |

22. Secondary Outcome: Maintenance Phase: Etrolizumab Serum Trough Concentration (for Arms/Timepoints Below LLOQ)
Description: As per protocol, the timepoints for each arm where more than a third of the samples were below the LLOQ only the Median and Max were reported.
Time Frame: Pre-dose (0 hour) at Baseline and Weeks 12, 24, 44, and 62
Population: All participants who received at least one dose of study drug, had evaluable PK data and were part of the timepoint that had more than a third of samples below LLOQ.
Measure: Median (Full Range); unit: micrograms per millilitre (μg/mL)
Arm/Group | Double-Blind Maintenance Phase: Placebo
Number analyzed (Participants) | 100
micrograms per millilitre (μg/mL)
  Week 12: number analyzed (Participants) | 0
  Week 24: number analyzed (Participants) | 76
  Week 24 | 0.0963 [NA to 1.89] — As per protocol, only the Median and Max were reported for timepoints where more than a third of the samples were LLOQ.
  Week 44: number analyzed (Participants) | 46
  Week 44 | 0.0400 [NA to 0.0400] — As per protocol, only the Median and Max were reported for timepoints where more than a third of the samples were LLOQ.
  Week 62: number analyzed (Participants) | 39
  Week 62 | 0.0400 [NA to 0.0400] — As per protocol, only the Median and Max were reported for timepoints where more than a third of the samples were LLOQ.

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 74
Arm/Group | Open-Label Induction Phase: Etrolizumab | Double-Blind Maintenance Phase: Etrolizumab | Double-Blind Maintenance Phase: Placebo
All-Cause Mortality (participants affected / at risk) | 0/358 | 0/108 | 0/102
Serious Adverse Events (participants affected / at risk) | 17/358 | 10/108 | 8/102
Other Adverse Events (participants affected / at risk) | 64/358 | 30/108 | 54/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Induction Phase: Etrolizumab (N=358) | Double-Blind Maintenance Phase: Etrolizumab (N=108) | Double-Blind Maintenance Phase: Placebo (N=102)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 6 (7) | 2 (2) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Induction Phase: Etrolizumab (N=358) | Double-Blind Maintenance Phase: Etrolizumab (N=108) | Double-Blind Maintenance Phase: Placebo (N=102)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 6 (9) | 9 (11)
Colitis ulcerative (Gastrointestinal disorders) | 24 (24) | 14 (16) | 34 (35)
Diarrhoea (Gastrointestinal disorders) | 5 (10) | 4 (4) | 8 (9)
Pyrexia (General disorders) | 8 (9) | 0 (0) | 6 (6)
Nasopharyngitis (Infections and infestations) | 22 (22) | 8 (10) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 8 (10) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT02165215/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT02165215/SAP_001.pdf